CLINICAL TRIAL: NCT00970346
Title: A Randomised, Double-blind, Placebo-controlled Dose-escalation Phase I Study to Evaluate the Safety and Tolerability of Inhaled Aerosolised OligoG CF-5/20 (G-block Oligosaccharide Derived From Alginate Polysaccharide) in Healthy Volunteers
Brief Title: Safety and Efficacy of Inhaled OligoG CF-5/20 for the Treatment Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AlgiPharma AS (Industry)
Collaborators: Smerud Medical Research International AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SMR-1916
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Cystic Fibrosis
Keywords: Digestive System Diseases; Genetic Diseases; Inborn; Respiratory Tract Diseases; Cystic Fibrosis; Lung Disease; Pancreatic Diseases
MeSH Terms: conditions — Cystic Fibrosis; Digestive System Diseases; Genetic Diseases, Inborn; Respiratory Tract Diseases; Lung Diseases; Pancreatic Diseases | interventions — oligoG CF-5-20

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhaled OligoG CF-5/20 (Experimental)
  Interventions: Drug: OligoG CF-5/20

INTERVENTIONS:
Drug: OligoG CF-5/20 — Inhaled OligoG CF-5/20 will be given to healthy volunteers with different concentrations to test tolerability of the drug

SUMMARY:
Cystic fibrosis (CF) is a disease caused by a mutation in the gene that makes the cystic fibrosis transmembrane regulator protein. As a result mucus stagnation, obstruction and plugging take place in the respiratory and gastrointestinal tract, the biliary and pancreatic duct, and in the reproductive system. The objective of this study is to determine the safety and tolerability of 3 days of daily dosing of OligoG CF-5/20 versus placebo in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male subjects aged 18 to 65 years inclusive
* Normal pulmonary function; i.e. FEV1 ≥ 80% of predicted (for age, sex, height and race) and FEV1/FVC ratio ≥ 0.7
* Subject's pre -study physical examination, vital signs and electrocardiogram (ECG) are normal or do not show any clinically significant abnormalities as determined by the investigator
* Subject's pre - study laboratory screen are normal or, if outside of the laboratory reference range, not considered clinically significant

Exclusion Criteria:

* History of any clinically relevant chronic respiratory disorder, including asthma
* Current smoker or smoked within the last 12 months
* History of significant drug or alcohol abuse (defined by the investigator). Subjects with a positive screen for alcohol or drugs of abuse at screening/admission will be excluded from participation in the study.
* Subject who has inhaled any drug in the last 30 days prior to Day 1
* Subject who has received one or more days of systemic pharmacological treatment in the 14 days immediately prior to Day 1
* Participation in a New Chemical Entity clinical study within the previous 16 weeks or a marketed drug clinical study within the previous 12 weeks
* Subjects with a clinically relevant history of significant hepatic, renal, endocrine, cardiac, nervous, psychiatric, gastrointestinal, pulmonary, haematological or metabolic disorder

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety and local tolerability of multiple dose administration of inhaled alginate oligosaccharide (OligoG CF-5/20) fragment in healthy volunteers, particular emphasis will be put on pulmonary functioning and pulmonary adverse events. | 3 days dosing

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Febbraro, Principal Investigator — Simbec Research
Locations (1):
- Merthyr Tydfil, United Kingdom